CLINICAL TRIAL: NCT02136485
Title: Mindfulness-based Stress Reduction in Multiple Sclerosis - a Randomised Controlled Trial
Brief Title: Mindfulness-based Stress Reduction in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GN14CH078
Record Dates: First submitted 2014-05-01; First posted 2014-05-13 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MBSR (Experimental): 8 weekly sessions each lasting 2.5 hours
  Interventions: Behavioral: Mindfulness-based stress reduction (MBSR)
- Control (Other): Control arm - waiting list control, once the intervention group has completed MBSR the control group will be invited to participate in MBSR
  Interventions: Other: waiting list control

INTERVENTIONS:
Behavioral: Mindfulness-based stress reduction (MBSR) — 8 sessions of MBSR
  Arms: MBSR
Other: waiting list control
  Arms: Control

SUMMARY:
This application concerns a proposed randomised controlled trial evaluating the use of Mindfulness-based stress reduction (MBSR) in people with Multiple Sclerosis (MS) in secondary care.

MS is an inherently stressful condition, and stress is thought to exacerbate MS. Mental health problems are common in MS, can impair quality of life, and lead to higher rates of suicide.

Prior research has shown that cognitive behavioural therapy (CBT) can help mitigate stress and diminish disease activity in MS, but effects are short-lived and there is thus a need to explore whether other psychological approaches might be more beneficial in this regard.

MBSR is another psychological stress reduction technique that is thought to operate differently to CBT, via cultivating a state of "meta-cognitive awareness" and has shown to be helpful when used in other long term conditions, such as chronic pain and anxiety, whilst Mindfulness-based cognitive therapy (MBCT - a derivative of MBSR) is effective in treating recurrent depression. All of these conditions are common in MS. However, mindfulness based interventions have not been well studied in MS.

The investigators propose to carry out a feasibility study to assess how acceptable and accessible MBSR is as a stress reduction technique in people with MS. The investigators would seek up to 50 participants who would then be randomly assigned to receive MBSR or their usual care. The investigators would seek measurements of health and wellbeing before, immediately following, and 3 months following the MBSR intervention. This would include basic demographic information (age, gender, ethnicity), measures of mental health, and physical health, as well as qualitative semi-structured interviews with selected participants. After this we would offer MBSR to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Having at baseline a Neurologist confirmed diagnosis of MS
* Can understand spoken and written English
* Score of less than or equal to 7 on the Expanded Disability Status Scale

Exclusion Criteria:

* Potentially life threatening physical or mental health comorbidities or conditions expected to significantly limit participation and adherence
* Current receipt of another form of psychological intervention (non-pharmacological)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-06-02 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Feasibility, accessibility, and acceptability of MBSR in people with MS | 5 months
  Completion rate

SECONDARY OUTCOMES:
Perceived stress symptoms (PSS) | 5 months
  PSS questionnaire
Health related Quality of Life | 5 months
  EuroQuol 5D (EQ-5D)
Multiple Sclerosis Quality of Life Inventory (MSQLI) | 5 months
  Measure of a) fatigue, b) chronic pain, c) sexual function, d) urinary function, e) bowel function, f) visual impairment, g) cognitive function, h) emotional distress

CONTACTS AND LOCATIONS:
Locations (1):
- NHS Centre for Integrative Care, Glasgow, United Kingdom

REFERENCES:
- [Derived] Simpson R, Simpson S, Wood K, Mercer SW, Mair FS. Using normalisation process theory to understand barriers and facilitators to implementing mindfulness-based stress reduction for people with multiple sclerosis. Chronic Illn. 2019 Dec;15(4):306-318. doi: 10.1177/1742395318769354. Epub 2018 Apr 26. No abstract available. PMID 29699410
- [Derived] Simpson R, Mair FS, Mercer SW. Mindfulness-based stress reduction for people with multiple sclerosis - a feasibility randomised controlled trial. BMC Neurol. 2017 May 16;17(1):94. doi: 10.1186/s12883-017-0880-8. PMID 28511703